CLINICAL TRIAL: NCT01811992
Title: A Non-randomized, Open-label Dose-finding Trial of Combined Cytotoxic and Immune-Stimulatory Strategy for the Treatment of Resectable Primary Malignant Glioma
Brief Title: Combined Cytotoxic and Immune-Stimulatory Therapy for Glioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: Phase One Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2015.024; HUM00057130 (Other: University of Michigan)
Record Dates: First submitted 2013-02-13; First posted 2013-03-15 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Malignant Glioma; Glioblastoma Multiforme
MeSH Terms: conditions — Glioma; Glioblastoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose escalation of Ad-hCMV-TK and Ad-hCMV-Flt3L (Experimental): This protocol is a dose escalation study of Ad-hCMV-TK and Ad-hCMV-Flt3L infused at the time of surgical resection followed by systemic oral administration of valacyclovir in addition to current standard of care with temozolomide and radiotherapy. Eligible subjects will be enrolled in six sequential dosing cohorts:
  * A= Ad-hCMV-TK: 1x10^10 vp and Ad-hCMV-Flt3L: 1x10^9 vp
  * B= Ad-hCMV-TK: 1x10^11 vp and Ad-hCMV-Flt3L: 1x10^9 vp
  * C= Ad-hCMV-TK: 1x10^10 vp and Ad-hCMV-Flt3L: 1x10^10 vp
  * D= Ad-hCMV-TK: 1x10^11 vp and Ad-hCMV-Flt3L: 1x10^10 vp
  * E= Ad-hCMV-TK: 1x10^10 vp and Ad-hCMV-Flt3L: 1x10^11 vp
  * F= Ad-hCMV-TK: 1x10^11 vp and Ad-hCMV-Flt3L: 1x10^11 vp
  Subjects will be treated sequentially with a minimum of 21 days before treatment of new subjects within a cohort or before dose escalation.
  Interventions: Biological: Dose Escalation of Ad-hCMV-TK and Ad-hCMV-Flt3L

INTERVENTIONS:
Biological: Dose Escalation of Ad-hCMV-TK and Ad-hCMV-Flt3L — Two adenoviral vectors will be used, each to deliver one of the therapeutic genes. Both vectors are human serotype 5, replication-defective, first generation adenoviral vectors deleted in E1a and E3 viral encoding regions. Each vector will constitutively express their respective therapeutic transgene (i.e. HSV1-TK or Flt3L) under the control of the human cytomegalovirus promoter (hCMV). Valacyclovir treatment will begin 1-3 days after vector administration at a dose of 2 grams given orally 3X per day for 14 days. A second course of valacyclovir will be given beginning Week 10.
  Radiation and chemotherapy will be administered as per standard of care.

SUMMARY:
Despite the marginal improvements in survival of patients suffering from malignant glioma treated with gene therapy vectors, the clinical trials conducted so far using viral vectors, in particular adenoviral vectors, have proven that the use of adenoviral vectors is a safe therapeutic approach, even in large, multicenter, phase 3 clinical trials. Treatment of malignant glioma using gene transfer modalities typically consists of surgical debulking of the tumor mass followed by the administration of the viral vectors into the brain tissue surrounding the tumor cavity. This study will combine direct tumor cell killing (TK) and immune-mediated stimulatory (Flt3L) gene transfer approaches delivered by first generation adenoviral vectors.

DETAILED DESCRIPTION:
This is a Phase 1, multiple center open label, dose escalation safety study of Ad-hCMV-TK and Ad-hCMV-Flt3L delivered to the peritumoral region after tumor resection. This study will combine direct tumor cell killing (TK) and immune-mediated stimulatory (Flt3L) gene transfer approaches delivered by first generation adenoviral vectors. Treatment with HSV1-TK is expected to kill transduced brain cells, thus exposing tumor antigen. Treatment with Flt3L, a cytokine known to cause proliferation of dendritic cells, should cause the migration of dendritic cells to the peritumoral brain and remaining tumor. There, they will be exposed to tumor antigens released from dying glioma cells through TK + valacyclovir-induced glioma cell death, and thus mediate a specific anti-malignant glioma immune response against remaining malignant glioma cells.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed supratentorial brain lesion compatible with a high grade glioma by MR (magnetic resonance) with no prior treatment with either gene therapy, chemotherapy or radiation treatments that is amenable to attempted gross total resection (GTR).Intraoperative histological frozen section at the time of tumor resection should be compatible with high-grade glioma. If intraoperative diagnosis is not high grade glioma, the patient will not be enrolled. "High grade glioma" can include:Glioblastoma multiforme (WHO grade IV); Anaplastic astrocytoma (WHO grade III); Anaplastic oligodendroglioma (WHO grade III); and Anaplastic ependymoma (WHO grade III).
* Karnofsky score ≥70 (Karnofsky scoring system used to quantify general well-being and activities of daily life; scores range from 0 to 100 where 100 represents perfect health and 0 represents death)
* CBC (complete blood count)/differential obtained within 14 days prior, with adequate bone marrow function defined as follows:
* Absolute neutrophil count (ANC) ≥ 1,500 cells/mm3;
* Platelets ≥ 100,000 cells/mm3;
* Hemoglobin ≥ 10.0 g/dl (Note: The use of transfusion or other intervention to achieve Hgb ≥10.0 g/dl is acceptable.);
* Adequate renal function, as defined below:
* BUN (blood urea nitrogen) ≤ 30 mg/dl within 14 days prior.
* Creatinine ≤ 1.7 mg/dl within 14 days prior.
* Adequate hepatic function, as defined below:
* Bilirubin ≤ 2.0 mg/dl within 14 days prior.
* ALT (alanine aminotransferase)/AST (aspartate aminotransferase) ≤ 3x laboratory upper limit of normal within 14 days prior.
* Male and female; both genders must use contraception if of reproductive capacity
* Capable of informed consent
* 18-75 years of age
* For women of child bearing age, a negative pregnancy test performed within 14 days of surgery

Exclusion Criteria:

* Diffusely multifocal lesion that is not amenable to GTR (gross total resection)
* Tumors infiltrating the cerebellum, bilateral corpus callosum ("butterfly glioma"), ventricular system, or brain stem
* Infratentorial high grade glioma
* Primary central nervous system (CNS) disease that would interfere with subject evaluation
* Current diagnosis of other cancer except curative cervical cancer in situ, basal or squamous cell carcinoma of the skin.
* Evidence of other significant disease including hematologic, renal or liver disease that is not explained by the patient's current medical condition or concomitant disease, (i.e. levels of absolute neutrophil count (ANC), hemoglobin, platelets, clotting time, serum creatinine, etc). Final decision on inclusion will be made by physician, concerning suitability of patient for surgery.
* HIV, Hepatitis B, Hepatitis
* Active systemic infection
* Immunosuppressive disorders (chronic steroid therapy, acquired or congenital immune deficiency syndromes, autoimmune disease)
* Serious medical conditions (CHF (congestive heart failure), angina, diabetes mellitus, Chronic obstructive pulmonary disease, abnormal bleeding diathesis)
* Any contraindication for undergoing MRI (magnetic resonance imaging)
* Pregnant or lactating females
* Unacceptable anesthesia risk
* Evidence of bleeding diathesis or use of anticoagulant medication or any medication that may increase the risk of bleeding that cannot be stopped prior to surgery.
* Prior gene therapy
* Allergy to valacyclovir or unable to take oral tablets

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 21 days post administration of study vectors
  Vectors AdhCMV- TK and Ad-hCMV-Flt3L were administered at time of surgery and the MTD determined by dose-limiting toxicities. Toxicities assessed and graded by the NCI Common Terminology Criteria for Adverse Events (CTCAE) v4.0.

SECONDARY OUTCOMES:
Number of Patients Alive at 12 and 24 Months | 24 Months
  To assess in a preliminary fashion the potential benefit of AdhCMV- TK and Ad-hCMV-Flt3L treatment of primary malignant gliomas by assessing overall survival (OS) at 12 and 24 months.

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Lowenstein, MD, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Health System Department of Neurosurgery, Ann Arbor, Michigan, United States

REFERENCES:
- [Result] Umemura Y, Orringer D, Junck L, Varela ML, West MEJ, Faisal SM, Comba A, Heth J, Sagher O, Leung D, Mammoser A, Hervey-Jumper S, Zamler D, Yadav VN, Dunn P, Al-Holou W, Hollon T, Kim MM, Wahl DR, Camelo-Piragua S, Lieberman AP, Venneti S, McKeever P, Lawrence T, Kurokawa R, Sagher K, Altshuler D, Zhao L, Muraszko K, Castro MG, Lowenstein PR. Combined cytotoxic and immune-stimulatory gene therapy for primary adult high-grade glioma: a phase 1, first-in-human trial. Lancet Oncol. 2023 Sep;24(9):1042-1052. doi: 10.1016/S1470-2045(23)00347-9. PMID 37657463
- [Derived] Lowenstein PR, Castro MG. Evolutionary basis of a new gene- and immune-therapeutic approach for the treatment of malignant brain tumors: from mice to clinical trials for glioma patients. Clin Immunol. 2018 Apr;189:43-51. doi: 10.1016/j.clim.2017.07.006. Epub 2017 Jul 15. PMID 28720549
- See also: Pubmed Link — https://pubmed.ncbi.nlm.nih.gov/37657463/